CLINICAL TRIAL: NCT04556435
Title: Analysis of Volatile Chemicals in the Breath of Lung Cancer Patients Using Infrared Spectroscopy
Brief Title: Breath Analysis in Early Stage Lung Cancer Using Infrared Spectroscopy
Status: Terminated | Type: Observational
Why Stopped: Change in the sponsor's business strategy (new focus on breast cancer)
Sponsor: Breathe BioMedical Inc (Industry)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-5606
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: Volatile Organic Compounds; Breath Analysis; Infrared Spectroscopy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LC Group: Participants will provide two breath samples by exhaling into the breath sampling apparatus and complete the Medical Questionnaire (medications, lifestyle, demographics, smoking history) and survey (lung health). Information related to LC diagnosis (histologic sub-type, tumor stage) will be collected.
- Control Group: Participants will provide two breath samples by exhaling into the breath sampling apparatus and complete the Medical Questionnaire (medications, lifestyle, demographics, smoking history) and survey (lung health).

SUMMARY:
The aim of this study is to sample and analyze volatile organic compounds (VOCs) from lung cancer patients and individuals without lung cancer ("healthy" controls). The breath sample analysis will help investigators describe and identify profiles of VOCs found in the breath of patients with lung cancer when compared to normal breath profiles using infrared spectroscopy. This work will help validate early proof of concept results conducted with prototype technology and later stage NSCLC breath samples, and inform future breath testing analysis.

DETAILED DESCRIPTION:
Globally, lung cancer accounts for the most cancer deaths in both sexes combined. It is believed to develop slowly through progressive accumulation of genetic mutations, hence the disease allows time for diagnosis and curative surgical treatment. Five year survival rates for non-small-cell lung carcinoma (NSCLC) can range from 57-61% when detected in the early stages of disease. This is compared with a survival rate of approximately 6% once distant metastases are present. However, disease diagnosis typically occurs when it has progressed to an advanced stage when patients present with signs and symptoms. Therefore, technologies capable of asymptomatic disease detection will significantly impact lung cancer specific mortality. Metabolomic profiling of cancer measures compounds produced as a result of cellular activity including volatile organic compounds (VOCs) in exhaled breath. Infrared spectroscopy is a proven technique for breath analysis that can measure chemical concentrations in the parts per trillion range for certain VOCs. When coupled with machine learning techniques, this has the potential to be a novel approach for disease detection using exhaled breath.

ELIGIBILITY:
Inclusion Criteria

LC Group:

* ≥ 18 years;
* Able to give informed consent;
* Eligible for lung cancer screening or lung cancer follow-up testing (biopsy, surgery);
* Clinical evidence of lung cancer (metastatic or primary), inclusive of those receiving non-curative treatment, has not yet been treated or is not currently on treatment;
* No history of or any other active cancer;
* Able to provide a breath sample;

Control Group:

* ≥ 18 years;
* Able to give informed consent;
* Eligible for lung cancer screening or lung cancer follow-up testing (biopsy, surgery);
* No history of lung cancer or any other active cancer and is eligible for lung cancer screening;
* Able to provide a breath sample;

Exclusion Criteria

* Has received or is currently receiving curative treatment and may no longer have lung cancer;
* Cannot give informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will analyze breath samples from study participants with diagnosed lung adenocarcinoma not currently receiving curative treatment and matched control participants without lung cancer. Prospective participants will be pre-screened prior to being approached about the study. Those scheduled for upcoming appointments will undergo a chart review to determine whether they meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
VOC spectral profile differences | 30 days after completion
  VOC spectral profiles will be compared between cohorts to identify statistical differences.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mahtabifard, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Mia Martinez, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Henderson B, Khodabakhsh A, Metsala M, Ventrillard I, Schmidt FM, Romanini D, Ritchie GAD, Te Lintel Hekkert S, Briot R, Risby T, Marczin N, Harren FJM, Cristescu SM. Laser spectroscopy for breath analysis: towards clinical implementation. Appl Phys B. 2018;124(8):161. doi: 10.1007/s00340-018-7030-x. Epub 2018 Jul 28. PMID 30956412
- See also: American Cancer Society. Cancer Facts & Figures 2019. — https://www.cancer.org/content/dam/cancer-org/research/cancer-facts-and-statistics/annual-cancer-facts-and-figures/2019/cancer-facts-and-figures-2019.pdf
- See also: American Cancer Society. Non-Small Cell Lung Cancer Survival Rates (2016) — https://www.cancer.org/cancer/lung-cancer/detection-diagnosis-staging/survival-rates.html